CLINICAL TRIAL: NCT03216447
Title: A Prospective, Multi-center, Open-labeled, Randomized Clinical Trial of Patient Adherence and Convenience to Immunosuppressive Agents in Newly Liver Transplant Recipients to Compare QD Early Conversion and BID Tacrolimus Formulation.
Brief Title: A Study of Patient Adherence and Convenience to Immunosuppressive Agents in Newly Liver Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Principal Investigator, Wei-Chen Lee, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201600495A3
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Liver Transplantation
Keywords: adherence; conversion; advagraf; prograf
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Masking Description: open labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Switch from Prograf to Advagraf on POD 15
  Interventions: Drug: Advagraf
- Control Arm (Active Comparator): Continue Prograf treatment
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Advagraf — Tacrolimus prolonged-release hard capsules (QD)
  Arms: Experimental Arm
Drug: Prograf — Tacolimus capsules (q12h)
  Arms: Control Arm

SUMMARY:
A study of patient adherence and convenience to immunosuppressive agents in newly liver transplant recipients - a prospective, multi-center, open-labeled, randomized clinical trial for comparison between once-daily early conversion and twice-daily tacrolimus formulation.

DETAILED DESCRIPTION:
This is prospective, multi-center, open-labeled, randomized study to investigate adherence of administration of once-daily tacrolimus formulation (Advagraf®) in newly Taiwanese (Chinese) liver transplant patients. The procedure of liver transplantation will follow the site-specific procedure. Each subject will be randomized on postoperative day 15 (POD15; defined Day 14 +/- 1)

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed and has signed an IRB approved informed consent form within 7 days (Day 7-13) prior to POD 15 and is willing and able to follow study procedure
* Patient is a primary liver transplant recipient
* Patient is 20 to 70 years of age
* Patient should be clearly conscious, fully understand and able to answer questionnaire

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a liver.
* Patient currently requires dialysis
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Patient has received a liver transplant from a non-heart beating donor
* Patient who is HCV negative has received an HCV positive (HCV RNA by PCR or HCV antibody) donor liver
* Patient who is HbsAg negative has received an HbsAg positive (HBV DNA by PCR or HBV antibody) donor liver
* Patient has received a liver transplant from a decrease donor > 70 years of age
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except hepatocellular carcinoma within UCSF Criteria and basal or non-metastatic squamous cell carcinoma of skin that has been treated successfully.
* Patient is hemodynamically unstable on POD 15

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence of administration of Advagraf in newly Taiwanese (Chinese) liver transplant patients. | Visit 1 (Day 14) to Visit 6 (Day 364) - 50 weeks observation
  • The adherence of enrolled 150 subjects will be assessed by the Basel assessment of adherence to immunosuppressive medications scale (BAASIS)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Lee, Principal Investigator — CGMH
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan